CLINICAL TRIAL: NCT03835013
Title: A Comparison of the Haemodynamic and Metabolic Effects of Intravenous Glucagon-like Peptide-1, Glucagon and Glucagon-like Peptide-1:Glucagon Co-agonism in Healthy Male Participants
Brief Title: Haemodynamic Effects of GLP-1 and Glucagon in Healthy Male Volunteers
Acronym: COCOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: COCOA; 18/EM/0417 (Other: REC-HRA); 250402 (Other: IRAS ID)
Record Dates: First submitted 2019-01-25; First posted 2019-02-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Sodium Chloride; Glucagon; Exenatide

STUDY DESIGN:
Intervention Model Description: Part A - 2 infusions Part B - 4 infusions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A - Infusion A (Placebo Comparator): 1. 60 minute intravenous infusion of 0.9% saline
     Followed by:
  2. 60 minute intravenous infusion of 0.9% saline
  Interventions: Drug: Saline 0.9%
- Part A - Infusion B (Active Comparator): 1. 60 minute intravenous infusion of glucagon 25ng/kg/min and 0.9% saline.
     Followed by:
  2. 60 minute infusion of glucagon 50ng/kg/min and 0.9% saline
  Interventions: Drug: Saline 0.9%; Drug: Glucagon (25ng/kg/min); Drug: Glucagon (50ng/kg/min)
- Part B - Infusion A (Active Comparator): A 60 minute intravenous infusion of 0.9% saline
  Interventions: Drug: Saline 0.9%
- Part B - Infusion B (Active Comparator): A 60 minute intravenous infusion of exenatide (50ng/min for 30 minutes followed by 25ng/min) and 0.9% saline
  Interventions: Drug: Saline 0.9%; Drug: Exenatide
- Part B - Infusion C (Active Comparator): A 60 minute intravenous infusion of glucagon (25ng/kg/min) and 0.9% saline
  Interventions: Drug: Saline 0.9%; Drug: Glucagon (25ng/kg/min)
- Part B - Infusion D (Active Comparator): A 60 minute intravenous infusion of exenatide (50ng/min for 30 minutes then 25ng/min) and glucagon (25ng/kg/min)
  Interventions: Drug: Glucagon (25ng/kg/min); Drug: Exenatide

INTERVENTIONS:
Drug: Saline 0.9% — Intravenous infusion of 0.9% saline
  Other Names: Placebo
  Arms: Part A - Infusion A; Part A - Infusion B; Part B - Infusion A; Part B - Infusion B; Part B - Infusion C
Drug: Glucagon (25ng/kg/min) — Intravenous infusion of glucagon 25ng/kg/min
  Other Names: Glucagon
  Arms: Part A - Infusion B; Part B - Infusion C; Part B - Infusion D
Drug: Glucagon (50ng/kg/min) — Intravenous infusion of glucagon 50ng/kg/min
  Other Names: Glucagon
  Arms: Part A - Infusion B
Drug: Exenatide — Intravenous infusion of Exenatide (loading 50ng/min for 30 minutes followed by 25ng/min for 30 minutes
  Arms: Part B - Infusion B; Part B - Infusion D

SUMMARY:
The study seeks to explore the cardiovascular effects of co-agonism at two peptide receptors, GLP-1 and glucagon. Glucagon, exenatide and 0.9% saline will be intravenously infused, both in isolation, and combination into healthy male participants. Overall, the aim of the study is to further our understanding on the role these endogenous substances play (both in isolation and combination) in haemodynamic regulation.

DETAILED DESCRIPTION:
Co-agonist peptides (such as at the GLP-1:glucagon receptor) are currently in clinical development for type 2 diabetes with the dual intention of reducing body weight and controlling blood glucose. However, there is a lack of data on the effects that co-agonism has on haemodynamic regulation.

Part A - Healthy male participants, by acting as their own control, will attend for two intravenous infusion visits (combination of 0.9% saline and glucagon). These will occur in a predefined but random order so that participants will be blinded to the infusion they are receiving. Each infusion visit will comprise of 15 minute baseline followed by a 120 minute infusion. Detailed non-invasive cardiovascular measurements (including peripheral/central blood pressure, heart rate, stroke volume, heart rate variability) and bloods (including insulin, glucose, GLP-1, glucagon) will be collected as part of the study. It was previously planned that GLP-1 7-36 amide 0.6pmol/kg/min and 1.2pmol/kg/min would be infused for Part A resulting in 5 infusions (rather than current 2 infusions). However due to supply/technical issues this was not possible and therefore exenatide (GLP-1 receptor agonist) shall be used in Part B.

Part B - Healthy male participants, by acting as their own control, will attend for four intravenous infusion visits (combination of 0.9% saline, glucagon, exenatide). These will occur in a predefined but random order so that participants will be blinded to the infusion they are receiving. Each infusion visit will comprise of 15 minute baseline followed by a 60 minute infusion. Detailed non-invasive cardiovascular measurements (including peripheral/central blood pressure, heart rate, stroke volume, heart rate variability) and bloods (including insulin, glucose, GLP-1, glucagon) will be collected as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* Aged 18 to 40
* Male
* Current non-smoker
* BMI >18.0 and <30kg/m2

Exclusion Criteria:

* Female
* Sustained Hypertension (sustained BP >160/100mmHg) or hypotension (systolic BP below 90 mmHg)
* Clinically significant heart disease
* Implanted heart pace-maker or implantable cardioverter defibrillator (ICD)
* Known active malignancy
* Known renal failure (creatinine >140μmol/L)
* Known diabetes mellitus (type 1 or 2)
* Use of vasoactive medications or NSAIDS/aspirin within 24 hours of study visits
* Use of formal anticoagulant therapy such as, but not limited to, heparin, warfarin or rivaroxaban
* Current involvement in the active treatment phase of other research studies, (excluding observations/noninterventional)
* Any other clinical reason which may preclude entry in the opinion of the investigator

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Heart rate (bpm)
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Brachial systolic and diastolic blood pressure (mmHg)
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Central systolic and diastolic blood pressure and mean arterial pressure (mmHg) measured with SphygmoCor XCEL
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Stroke volume (ml) measured by bioimpedance
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Cardiac output (L/min) measured by bioimpedance
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  peripheral vascular resistance (dynes/sec/cm)
Changes in haemodynamic parameters following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Heart rate variability (normalised low frequency, LF, high frequency, HF and LF/HF ratio)

SECONDARY OUTCOMES:
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-5 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Glucose, in mmol/L
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  C-peptide, in pmol/L
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Glucagon, in pg/ml
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Insulin, in pmol/L
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Free fatty acids, in μmol/L
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Total GLP-1 and total active GLP-1, in pg/ml
Changes in glucose homeostasis following intravenous infusion of 0.9% saline, glucagon, exenatide and their combination. | Comparison between 2 hour infusion visit 1-2 (Part A) / 1 hour infusion visit 1-4 (Part B), over a maximum period of 15 weeks
  Gastric inhibitory polypeptide, in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, MA DM FRCP, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom